CLINICAL TRIAL: NCT07379957
Title: Imlifidase for Highly Sensitized Kidney Transplant Recipients With a posItive crossmAtch Against a Deceased Donor: Results of Kidney Transplantations Performed in Accordance to the French Guidelines.
Acronym: ISKIA
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX2025/031
Record Dates: First submitted 2025-09-26; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Kidney Transplantation
Keywords: End-stage renal disease; kidney transplant rejection; recombinant cysteine protease derived from Streptococcus pyogenes; imlifidase
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient eligible for Imlifidase
- Patient eligible for imlifidase and transplanted with
- Patient eligible for imlifidase but transplanted without

SUMMARY:
Imlifidase is a recombinant cysteine protease derived from Streptococcus pyogenes and produced in Escherichia coli, which has the ability to cleave and degrade all human IgGs. Four to six hours after imlifidase infusion, the entire IgG pool is degraded into F(ab')2 and Fc fragments. In vitro, imlifidase inhibits HLA antibody-mediated NK cell activation and antibody-dependent cell-mediated cytotoxicity. Imlifidase degrades also the IgG of the B cell Receptor (BCR), inhibiting BCR-mediated cell signal, transiently preventing memory B cell response to antigenic stimulation and their transition into antibody-producing cells.

Two clinical studies have been designed to determine whether imlifidase could inactivate IgG donor-specific antibodies as a desensitization strategy in highly sensitized candidates for kidney transplantation. In the phase I/II study, 25 patients were transplanted in Sweden and United States. Among them, 18 had a positive flow cytometry crossmatch (FCXM) and 2 a positive complement-dependent cytotoxicity crossmatch (CDCXM). In the phase II study (Highdes Trial), 19 patients with an incompatible living or deceased donor from the United States, Sweden, and France were included. Among them, 7, 18, 2, and 8 had respectively a positive T-cell FCXM, positive B-cell FCXM, positive T-cell CDCXM, and positive B-cell CDCCXM. The primary efficacy endpoint was the ability of Imlifidase to convert a positive XM to a negative one. Conversion of baseline positive XM to negative within 24 h after Imlifidase treatment occurred in 89.5% (n=17) of the 19 patients. In the follow-up study including all the patients transplanted after Imlifidase desensitization, the antibody-mediated rejection rate (AMR) was at 39%, most of them occurring during the first month post-transplantation. Three-year death-censored graft survival was 93% in patients with AMR and 77% in the others. Three-year patient survival was 85% in patients with AMR and 94% in the others. No safety signal was reported.

Based on these data, Imlifidase is now indicated as a desensitization agent of highly sensitized adult kidney transplant patients with positive crossmatch against an available ABO-compatible deceased donor. It should be reserved for patients unlikely to be transplanted under the available kidney allocation system including the prioritization program for highly sensitized patients (https://www.ema.europa.eu). Therefore, the French Society of Transplantation (SFT), the French-speaking Society of Nephrology, Dialysis and Transplantation (SFNDT) and the French Society of Histocompatibility and Immunogenetics (SFHI) have proposed French recommendations for patient selection, choice of antibodies characteristics, treatment and follow-up in order to homogenize practices.

Although this new treatment addressed an unmet medical need, its authorization was based on only two small-scale studies. Therefore, additional data on long-term graft function and survival are required in patients treated by imlifidase.

DETAILED DESCRIPTION:
Kidney transplantation is the treatment of choice for patients with end-stage renal disease. However, highly sensitized patients have a very difficult access to transplantation because of a very low number of compatible donors. Imlifidase is a major breakthrough in kidney transplantation, because it allows transplanting these highly sensitized patients considered as untransplantable until now. The findings coming from the ISKIA study will help to refine the use and implementation of imlifidase in this population.

The main objective of this retrospective study is to analyze the efficacy and safety of kidney transplantations performed with a positive crossmatch against a deceased donor, where imlifidase is used in accordance to the French guidelines.

The secondary objectives of the ISKIA study are:

* To identify the characteristics and analyze the outcome of kidney recipients eligible to imlifidase but transplanted without imlifidase
* To identify the characteristics of kidney recipients eligible to imlifidase but not transplanted

ELIGIBILITY:
Inclusion Criteria:

* Highly sensitized adult kidney transplant candidates
* Eligible to imlifidase (patient with a delisting of at least one A, B, DR, DQ HLA antibody)

Exclusion Criteria:

* Age < 18 years-old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: When a kidney transplant candidate eligible to imlifidase is identified in a transplant center in France, HLA antibodies are delisted by the HLA laboratory, according to the French guidelines. Following this delisting, the patients can be transplanted with or without imlifidase or stay on dialysis.
  Bordeaux University Hospital will establish agreements with the 20 other university hospitals who have patients eligible to imlifidase.
  An implementation visit will be carried out at each CHU to:
  1. identify patients already eligible for imlifidase,
  2. set up a system to inform the Bordeaux CHU, as the coordinating center, when new incident patients eligible for imlifidase are identified,
  3. offer all identified patients' inclusion in the ISKIA study
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of transplantations performed with or without imlifidase among the eligible patients | Year 1, year 2 and year 3 after kidney transplantation
  CRISTAL register

SECONDARY OUTCOMES:
Incidence of HLA donor-specific antibodies (DSA) rebound after transplantation | Days 3, 5, 7, 10, and month 1, month 3 and month 12, after kidney transplantation
  DSA analysis on a Luminex platform
Timing of HLA donor-specific antibodies (DSA) rebound after transplantation | Days 3, 5, 7, 10, and month 1, month 3 and month 12, after kidney transplantation
  DSA analysis on a Luminex platform
Incidence of antibody-mediated rejection | Day 10, month 3 and month 12 after kidney tranplantation
  Protocol and indication biopsies
eGFR | Days 7, 14, month 1, month 3 and month 12 after kidney transplantation
  Estimated eGFD based on serum creatinine (CKD-epi formula)
Description of infection on post-transplantation | Year 1, year 2 and year 3 after kidney transplantation
  Collection of events on patients' records
Description of cancer post-transplantation | Year 1, year 2 and year 3 after kidney transplantation
  Collection of events on patients' records concerning cancer onset post-transplantation
Patient and graft survivals | Year 1, year 2 and year 3 after kidney transplantation
  Collection of events on patients' records concerning graft survivals
Patients placed on the waiting list after transplantation | Year 1, year 2 and year 3 after kidney transplantation
  Patients placed on the waiting list after transplantation will be estimated thanks to CRISTAL register

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - CHU Amiens Picardie Site Sud, Amiens
  - Hôpital de Bois-Guillaume, Bois-Guillaume
  - Hôpital Pellegrin, Bordeaux
  - CHU Caen Normandie, Caen
  - Hôpital Henri Mondor, Créteil
  - CHU de Grenoble Alpes, Grenoble
  - Hôpital Huriez, Lille
  - Hôpital Edouard Herriot, Lyon
  - Hôpital de la Conception, Marseille
  - CHU de Nantes, Nantes
  - Hôpital Pasteur, Nice
  - Hôpital Bicêtre, Paris
  - Hôpital Necker, Paris
  - Hôpital Saint-Louis, Paris
  - CHU de Reims, Reims
  - CHU Saint Etienne, Saint-Etienne
  - CHU de Strasbourg, Strasbourg
  - Hôpital Foch, Suresnes
  - Hôpital Rangueil, Toulouse
  - CHU Tours Bretonneau, Tours